CLINICAL TRIAL: NCT00311558
Title: Phase I Evaluation of Sodium Stibogluconate in Combination With Interferon α-2b for Solid Tumors, Lymphoma or Myeloma
Brief Title: Sodium Stibogluconate and Interferon in Treating Patients With Advanced Solid Tumors, Lymphoma, or Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE-CCF-7059; P30CA043703 (NIH); CASE-CCF-7509 (Other: IRB number); CASE-CCF-1062 (Other: IRB number); CASE 2Y06 (Other: IRB Number)
Record Dates: First submitted 2006-04-05; First posted 2006-04-06 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Cancer
Keywords: stage IV melanoma; stage IV adult soft tissue sarcoma; recurrent melanoma
MeSH Terms: conditions — Neoplasms; Melanoma; Sarcoma | interventions — Introns; Antimony Sodium Gluconate; Interferons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SSG & INF (Experimental): 1 arm study: SSG & interferon
  Interventions: Biological: recombinant interferon alfa-2b; Drug: sodium stibogluconate; Drug: SSG & interferon

INTERVENTIONS:
Biological: recombinant interferon alfa-2b — SSG x 5 week
  Other Names: Sodium Stibocluconate
Drug: sodium stibogluconate — SSG & IFN
Drug: SSG & interferon — 1 arm study with SSG & interferon
  Other Names: Sodium Stiboglucante

SUMMARY:
RATIONALE: Sodium stibogluconate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Interferon may interfere with the growth of cancer cells. Giving sodium stibogluconate together with interferon may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of sodium stibogluconate when given together with interferon in treating patients with advanced solid tumors, lymphoma, or myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Confirm the tolerance, safety, and maximum tolerated dose of sodium stibogluconate (SSG) in combination with interferon alfa-2b in patients with advanced solid tumors, lymphoma, or myeloma.

Secondary

* Quantify the effect of SSG on interferon alfa-2b-induced gene modulation and signal transduction pathways by measurement of the serum-soluble gene products β-2 microglobulin, immune serum globulin 15, and neopterin.
* Define the effectiveness of SSG in inhibiting the protein tyrosine phosphatases src homology proteins (SHP)-1 and SHP-2 assayed from peripheral blood leukocytes of patients receiving SSG in combination with interferon alfa-2b.
* Define pharmacokinetics of SSG in serum at escalating doses.
* Assess clinical response to the combination of SSG and interferon alfa-2b.

OUTLINE: This is an open-label, dose-escalation study of sodium stibogluconate (SSG).

Patients receive SSG IV over 15 minutes on days 1, 15-19, and 22-26 and interferon alfa-2b subcutaneously daily on days 8-12 and 15-28. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 6 patients receive escalating doses of SSG until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignancy, including, but not limited to, any of the following:

  * Renal cell carcinoma
  * Melanoma
  * Kaposi's sarcoma
  * Breast, prostate, colorectal, or lung adenocarcinoma
  * Bone and soft tissue sarcomas
  * Lymphoma
  * Myeloma
  * Tumors of neuroendocrine and endothelial cell origin
* Stage IV disease
* Refractory disease, resistant to established treatments, or no effective treatment available
* Measurable or evaluable disease
* CNS metastases allowed if no prior definitive therapy within the past 3 months and no glucocorticoids required

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Granulocyte count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Creatinine < 1.0 times upper limit of normal (ULN)
* Creatinine clearance ≥ 60 mL/min
* Bilirubin < 1.5 times ULN
* AST/ALT < 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* No history of any of the following:

  * Atrial fibrillation, atrial flutter, or other serious arrhythmia (excluding asymptomatic atrial and ventricular premature complexes)
  * Congestive heart failure currently requiring treatment
  * Angina pectoris
  * Other severe cardiovascular disease (i.e., New York Heart Association class III or IV heart disease)
* No baseline ECG abnormalities suggestive of cardiac conduction delay, i.e., 1° or greater atrio-ventricular block and/or complete or incomplete (QRS > 120 ms) bundle branch block, or repolarization abnormalities (i.e., QTc ≥ 0.48 sec)
* No systemic infections requiring antibiotics within the past 14 days
* No known hepatitis B surface antigen positivity
* Psychologically prepared to participate in study treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 weeks since prior interferon (IFN) therapy and/or ≤ 400 million units of IFN
* At least 3 weeks since prior major surgery
* At least 3 weeks since prior radiation therapy or chemotherapy
* No prior solid organ allografts or allogeneic bone marrow transplantation
* No concurrent daily glucocorticoids except for physiological replacement
* No other concurrent medications known to prolong QT interval

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-10; Primary Completion 2011-05 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Tolerance, safety, and maximum tolerated dose at 1 week after each course | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ernest C. Borden, MD, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio, United States